CLINICAL TRIAL: NCT04578834
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase III Study to Evaluate the Efficacy and Safety of LNP023 in Primary IgA Nephropathy Patients
Brief Title: Study of Efficacy and Safety of LNP023 in Primary IgA Nephropathy Patients
Acronym: APPLAUSE-IgAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLNP023A2301
Record Dates: First submitted 2020-09-09; First posted 2020-10-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: IgA Nephropathy
Keywords: LNP023; IgA nephropathy; IgAN, proteinuria; UPCR; eGFR; eGFR slope; kidney function decline
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria | interventions — iptacopan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LNP023 200mg b.i.d (Experimental)
  Interventions: Drug: LNP023
- Placebo to LNP023 200mg b.i.d (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo to LNP023 200mg b.i.d
  Arms: Placebo to LNP023 200mg b.i.d
Drug: LNP023 — LNP023 200mg b.i.d
  Other Names: iptacopan
  Arms: LNP023 200mg b.i.d

SUMMARY:
The study is designed as a multicenter, randomized, double-blind, placebo controlled study to demonstrate the superiority of iptacopan (LNP023) at a dose of 200 mg b.i.d. compared to placebo on top of maximally tolerated ACEi or ARB on reduction of proteinuria and slowing renal disease progression in primary IgA Nephropathy patients.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy and safety of iptacopan (LNP023) compared to placebo on proteinuria reduction and slowing disease progression in primary IgAN patients. The study will be the pivotal trial for registration of LNP023 in IgA Nephropathy patients with the aim to demonstrate a clinically meaningful reduction in proteinuria by LNP023 vs. placebo as assessed by reduction in urine protein to creatinine ratio (UPCR) sampled from a 24 hour urine collection at an IA at 9 months. The trial will continue in a blinded fashion to confirm long-term efficacy based on annualized total slope of eGFR decline over 24 months to provide confirmatory evidence of LNP023 efficacy and safety in treating patients with IgAN. The trial will enroll approximately 470 participants; 430 biopsy-proven IgAN participants with eGFR ≥30 mL /min/1.73m2 (main study population) and up to approximately 40 participants with eGFR 20 to <30 mL/min/1.73m2 (severe renal impairment (SRI) population).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years of age with an eGFR level and biopsy-confirmed IgA nephropathy as follows:
* For patients eGFR* ≥ 45ml/min/1.73m2, a qualifying biopsy performed within the last 5 years is required.
* For patients with eGFR* 30 to <45ml/min/1.73m2, a qualifying biopsy performed within 2 years with < 50% tubulointerstitial fibrosis is required.
* For patients with eGFR* 20 to <30ml/min/1.73m2, a qualifying biopsy performed at any time.

In all cases, if a historical biopsy is not available, one may be performed during screening. *eGFR calculated using the CKD-EPI formula (or modified MDRD formula according to specific ethnic groups and local practice guidelines)

* Proteinuria due to primary diagnosis of IgA nephropathy as assessed at screening by UPCR ≥1 g/g (113 mg/mmol) sampled from FMV or 24h urine collection, as well as at the completion of the run-in period by UPCR ≥1 g/g (113 mg/mmol) calculated as the (geometric) mean of two 24h urine collections obtained within 14 days of each other at baseline.
* Vaccination against Neisseria meningitidis and Streptococcus pneumoniae infection is required prior to the start of study treatment. If the patient has not been previously vaccinated, or if a booster is required, vaccine should be given according to local regulations at least 2 weeks prior to first study drug administration. If study treatment has to start earlier than 2 weeks post vaccination, prophylactic antibiotic treatment should be initiated.
* If not previously vaccinated, vaccination against Haemophilus influenzae infections should be given, if available and according to local regulations, at least 2 weeks prior to first study drug administration.
* All patients must have been on supportive care including stable dose regimen of ACEi or ARB at either the locally approved maximal daily dose or the maximally tolerated dose (per investigators' judgment) for approximately 90 days before first study drug administration. In addition, if patients are taking diuretics, other antihypertensive medication, or other background medication for IgAN, the doses should also be stabilized for approximately 90 days prior to the first dosing of study treatment.

Exclusion Criteria:

* Any secondary IgAN as defined by the investigator; secondary IgAN can be associated with cirrhosis, celiac disease, Human Immunodeficiency Virus (HIV) infection, dermatitis herpetiformis, seronegative arthritis, small-cell carcinoma, lymphoma, disseminated tuberculosis, bronchiolitis obliterans, and inflammatory bowel disease, familial mediterranean fever, etc.
* Sitting office SBP >140 mmHg or DBP >90 mmHg at the randomization visit
* Patients previously treated with immunosuppressive or other immunomodulatory agents such as but not limited to cyclophosphamide, rituximab, infliximab, eculizumab, canakinumab, mycophenolate mofetil (MMF) or mycophenolate sodium (MPS), cyclosporine, tacrolimus, sirolimus, everolimus, or systemic corticosteroids exposure (>7.5 mg/d prednisone/prednisolone equivalent) within 90 days (or 180 days for rituximab) prior to first study drug administration. Participants previously or currently treated with oral budesonide. Participants treated with endothelin (receptor) antagonists within 90 days prior to first study drug administration.
* Prior use of iptacopan (LNP023) or prior enrollment in any other LNP023 clinical trial where study drug was taken, including matching placebo
* History of recurrent invasive infections caused by encapsulated organisms, such as meningococcus and pneumococcus.
* Active systemic bacterial, viral (including COVID-19) or fungal infection within 14 days prior to study drug administration.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Ratio to baseline in Urine Protein to Creatinine Ratio (sampled from 24h urine collection) at 9 months | Baseline and 9 months
  Evaluated at interim analysis - To demonstrate superiority of LNP023 vs. placebo in the change of proteinuria at 9 months by measuring Urine Protein to Creatinine Ratio sampled from a 24h urine collection.
Annualized total estimated Glomerular Filtration Rate (eGFR) slope over 24 months). | Baseline and 24 months
  Evaluated at the final analysis - to demonstrate superiority of LNP023 vs. placebo in slowing IgAN progression measured by the annualized total slope of Estimated Glomerular Filtration Rate (eGFR) change over 24 months.

SECONDARY OUTCOMES:
Change from baseline in estimated glomerular filtration rate at 9 months | Baseline and 9 months
  Evaluated at interim analysis - To evaluate the effect of LNP023 vs. placebo on slowing estimated glomerular filtration rate decrease as measured by the change from baseline in eGFR
Proportion of participants reaching Urine Protein To Creatinine Ratio <1g/g without receiving Corticosteroids/Immunosuppressant or other newly approved drugs or initiating new background therapy for treatment of IgAN or Kidney Replacement Therapy (KRT) | Baseline and 9 months
  Evaluated at interim analysis - To assess the effect of LNP023 vs. placebo on the proportion of study participants reaching proteinuria below 1g/g of Urine Protein To Creatinine Ratio (sampled from 24h urine collection) at 9 months.
Annualized total Estimated Glomerular Filtration Rate slope estimated over 12 months | Baseline and 12 months
  Evaluated at interim analysis - To evaluate the effect of LNP023 vs. placebo on slowing IgAN progression measured by the annualized total slope of Estimated Glomerular Filtration Rate change over 1 year.
Change from baseline to 9 months in the fatigue scale measured by the Functional Assessment Of Chronic Illness Therapy-Fatigue questionnaire | Baseline and 9 months
  Evaluated at interim analysis - To assess the effect of LNP023 vs. placebo on the change from baseline to 9 months in fatigue scale measured by the Functional Assessment Of Chronic Illness Therapy-Fatigue questionnaire.
Time from randomization to first occurrence of composite kidney failure endpoint event | Up to 24 months
  Evaluated at final analysis - demonstrate the superiority of LNP023 vs. placebo on delaying the time to first occurrence of a composite kidney failure endpoint, defined as reaching either sustained ≥30% decline in Estimated Glomerular Filtration Rate (eGFR) relative to baseline or sustained eGFR <15 mL/min/1.73m2 or maintenance dialysis or receipt of kidney transplant or death from kidney failure.
Ratio to baseline in Urine Protein-To-Creatinine Ratio (sampled from 24h urine collection) at 9 months | Baseline and 9 months
  Evaluated at final analysis - To demonstrate superiority of LNP023 vs. placebo in the change of proteinuria at 9 months by measuring Urine Protein To Creatinine Ratio sampled from a 24h urine collection.
Proportion of participants reaching Urine Protein-To-Creatinine Ratio <1g/g without receiving Corticosteroids/Immunosuppressant Therapy or other newly approved drugs or initiating new background therapy for treatment of IgAN or initiating KRT | Baseline and 9 months
  Evaluated at final analysis - To demonstrate the superiority of LNP023 vs. placebo on the proportion of study participants reaching proteinuria below 1g/g of Urine Protein To Creatinine Ratio (sampled from 24h urine collection) at 9 months.
Change from baseline to 9 months in the fatigue scale measured by the Functional Assessment Of Chronic Illness Therapy-Fatigue questionnaire. | Baseline and 9 months
  Evaluated at final analysis - To demonstrate the superiority of LNP023 vs. placebo on the change from baseline to 9 months in the fatigue scale measured by Functional Assessment Of Chronic Illness Therapy-Fatigue questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (157):
- United States (22):
  - AZ Kidney Dise and Hypertension Ctr, Glendale, Arizona
  - AKDHC Medical Research ServicesLLC, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - Kaiser Permanente, San Diego, California
  - North America Research Institute, San Dimas, California
  - University of Colorado Anschutz, Aurora, Colorado
  - Nephrology Associates PA, Newark, Delaware
  - Boise Kidney and Hypertension, Boise, Idaho
  - CaRe Research, Chubbuck, Idaho
  - Nep Assoc of Northern Illinois, Hinsdale, Illinois
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Womens Hosp Harvard Med School, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Clin Rsrch Consult a JCCT Company, Kansas City, Missouri
  - DaVita Clinical Research, Las Vegas, Nevada
  - New Jersey Kidney Care, Jersey City, New Jersey
  - Columbia University Irving Medical, New York, New York
  - Dallas Renal Group, Dallas, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Univ of Washington Medi Cen, Seattle, Washington
- Argentina (3):
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Santa Fe
- Australia (5):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, St Albans, Victoria
- Belgium (3):
  - Novartis Investigative Site, Roeselare, West-Vlaanderen
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Leuven
- Brazil (5):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Sao Jose Rio Preto
- Novartis Investigative Site, Oshawa, Ontario, Canada
- Novartis Investigative Site, Temuco, Chile
- China (20):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Luoyang, Henan
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Yinchuan, Ningxia
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Ningbo, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Ningbo
  - Novartis Investigative Site, Qingdao
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Shenzhen
- Colombia (2):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
- Novartis Investigative Site, Prague, Czechia
- Denmark (4):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Arhus N
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Odense C
- France (3):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
- Germany (13):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
- Hungary (3):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Szeged
- India (3):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Hyderabad, Telangana
- Israel (3):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
- Italy (2):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Napoli
- Japan (15):
  - Novartis Investigative Site, Kasugai, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Toyota, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Ōmihachiman, Shiga
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
- Malaysia (2):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (3):
  - Novartis Investigative Site, Mexicali, Baja California Norte
  - Novartis Investigative Site, Mexico City
  - Novartis Investigative Site, Querétaro
- Novartis Investigative Site, Groningen, Provincie Groningen, Netherlands
- Norway (2):
  - Novartis Investigative Site, Nordbyhagen, Oslo County
  - Novartis Investigative Site, Bergen
- Russia (3):
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Košice, Slovakia, Slovakia
- Slovenia (2):
  - Novartis Investigative Site, Maribor, Slovenia
  - Novartis Investigative Site, Ljubljana
- Novartis Investigative Site, Bloemfontein, Free State, South Africa
- South Korea (6):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu
- Spain (4):
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Seville
- Sweden (2):
  - Novartis Investigative Site, Danderyd
  - Novartis Investigative Site, Stockholm
- Taiwan (5):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, New Taipei City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (8):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Köseköy, Kocaeli
  - Novartis Investigative Site, Antalya, Konyaalti
  - Novartis Investigative Site, Kayseri, Melikgazi
  - Novartis Investigative Site, Istanbul, Sariyer
  - Novartis Investigative Site, Istanbul, Sultangazi
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Mersin, Yenisehir
- United Kingdom (4):
  - Novartis Investigative Site, Newcastle upon Tyne, Tyne and Wear
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Salford
- Vietnam (2):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Perkovic V, Barratt J, Rovin B, Kashihara N, Maes B, Zhang H, Trimarchi H, Kollins D, Papachristofi O, Jacinto-Sanders S, Merkel T, Guerard N, Renfurm R, Hach T, Rizk DV; APPLAUSE-IgAN Investigators. Alternative Complement Pathway Inhibition with Iptacopan in IgA Nephropathy. N Engl J Med. 2025 Feb 6;392(6):531-543. doi: 10.1056/NEJMoa2410316. Epub 2024 Oct 25. PMID 39453772
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] Zhang H, Rizk DV, Perkovic V, Maes B, Kashihara N, Rovin B, Trimarchi H, Sprangers B, Meier M, Kollins D, Papachristofi O, Milojevic J, Junge G, Nidamarthy PK, Charney A, Barratt J. Results of a randomized double-blind placebo-controlled Phase 2 study propose iptacopan as an alternative complement pathway inhibitor for IgA nephropathy. Kidney Int. 2024 Jan;105(1):189-199. doi: 10.1016/j.kint.2023.09.027. Epub 2023 Oct 31. PMID 37914086
- [Derived] El Karoui K, Fervenza FC, De Vriese AS. Treatment of IgA Nephropathy: A Rapidly Evolving Field. J Am Soc Nephrol. 2024 Jan 1;35(1):103-116. doi: 10.1681/ASN.0000000000000242. Epub 2023 Sep 29. PMID 37772889
- [Derived] Reich HN, Floege J. How I Treat IgA Nephropathy. Clin J Am Soc Nephrol. 2022 Aug;17(8):1243-1246. doi: 10.2215/CJN.02710322. Epub 2022 Jun 8. No abstract available. PMID 35675911